CLINICAL TRIAL: NCT06517550
Title: Effect of Protective Lung Ventilation Measures on Pulmonary Complications in Elderly Patients After Upper Abdominal Laparoscopy
Brief Title: Pulmonary Complications in Elderly Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: China-Japan Friendship Hospital (Other)
Responsible Party: Principal Investigator, Jinjing Zhang, Principal Investigator, China-Japan Friendship Hospital
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: 2021-HX-54
Record Dates: First submitted 2024-07-19; First posted 2024-07-24 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2024-10

CONDITIONS: Postoperative Complications
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PEEP 5 cmH2O (No Intervention): During the surgical mechanical ventilation process, a constant PEEP value of 5 cmH2O is set.
- Personalized PEEP (Experimental): During surgical mechanical ventilation, individualized PEEP values are set based on each patient's lung condition.
  Interventions: Other: positive end-expiratory pressure while mechanical ventilation

INTERVENTIONS:
Other: positive end-expiratory pressure while mechanical ventilation — a parameter in ventilator
  Arms: Personalized PEEP

SUMMARY:
The incidence of postoperative pulmonary complications in elderly patients undergoing upper abdominal laparoscopic surgery remains high, and the lung protective mechanical ventilation strategy aims to reduce the incidence of lung injury caused by ventilators. PEEP, as an important protective ventilation strategy, maintains end expiratory alveolar volume to improve intraoperative oxygenation and pulmonary respiratory mechanics, and plays a protective role in the lungs; Personalized PEEP is the most beneficial, especially for elderly patients. However, there is currently no ideal way to achieve precise and personalized regulation of PEEP. This project aims to target and control intraoperative mechanical ventilation to drive pressure, personalize PEEP titration, and conduct a randomized controlled study on perioperative changes in pulmonary oxygenation function and pulmonary complications in elderly patients undergoing upper abdominal laparoscopy.

ELIGIBILITY:
Inclusion Criteria:

* ASA<III、 general anesthesia, 60-80 years, BMI<30kg/m2, pneumoperitoneum time>0.5h, laparoscopic surgery on the upper abdomen (stomach, liver, gallbladder)

Exclusion Criteria:

* Severe anemia (Hb<60g/L), OSA, severe COPD (FEV1<30% pre), asthma, bronchiectasis, preoperative pulmonary infection, respiratory failure, thoracic deformity, postoperative return to ICU, heart function grade III-IV, severe liver and kidney dysfunction (Child B or C, dialysis), intraoperative bleeding greater than 30% of blood volume.

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-11-01 (Actual)

PRIMARY OUTCOMES:
the changes of oxygenation index | pre-surgery, leave-PACU, one-day after surgery and 7-day after surgery
  The patients' changes of Oxygenation index when leave-PACU, one-day after surgery and 7-day after surgery compared with pre-sugery oxygenation index

SECONDARY OUTCOMES:
Incidence of pulmonary complications | 30 and 90 days after surgery
  Incidence of pulmonary complications at 30 and 90 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Feng X Ren, doctor, Principal Investigator — China-Janpan Friendship Hospital
Locations (1):
- China-Japan Friendship Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF, CSR
Time Frame: two years after the research and they will be available forever
Access Criteria: all researchers